CLINICAL TRIAL: NCT00044291
Title: Phase III Study of Atamestane Plus Toremifene Versus Letrozole in Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Biomed 777-CLP-29
Record Dates: First submitted 2002-08-23; First posted 2002-08-27 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Breast Neoplasms; Neoplasms, Hormone-dependent
Keywords: Atamestane; Toremifene; Letrozole; Aromatase inhibitor; Receptor-positive; First line therapy; Estrogen blocker; Metastatic breast cancer; Locally advanced breast cancer; Locally recurrent breast cancer; stage IV breast cancer; ductal breast carcinoma; lobular breast carcinoma; stage IIIA breast cancer; stage IIIB breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms, Hormone-Dependent; Carcinoma, Ductal, Breast; Carcinoma, Lobular | interventions — atamestane; Toremifene; Letrozole; Aromatase Inhibitors; Estrogen Receptor Modulators

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Atamestane + toremifene (Experimental)
  Interventions: Drug: atamestane; Drug: toremifene; Drug: aromatase inhibition; Procedure: hormone therapy; Procedure: endocrine therapy; Procedure: antiestrogen therapy
- Letrozole + placebo (Active Comparator)
  Interventions: Drug: letrozole; Drug: aromatase inhibition; Procedure: hormone therapy; Procedure: endocrine therapy

INTERVENTIONS:
Drug: atamestane
  Arms: Atamestane + toremifene
Drug: toremifene
  Arms: Atamestane + toremifene
Drug: letrozole
  Arms: Letrozole + placebo
Drug: aromatase inhibition
Procedure: hormone therapy
Procedure: endocrine therapy
Procedure: antiestrogen therapy
  Arms: Atamestane + toremifene

SUMMARY:
The purpose of this study is to determine whether the first line combination hormonal therapy of an experimental drug, atamestane, plus an FDA-approved drug, toremifene (Fareston®), is more effective than another approved drug, letrozole (Femara®), in delaying the growth of breast cancer in postmenopausal patients with locally advanced or metastatic breast cancer, and whether the side effects of the combination are different from the side effects of letrozole.

DETAILED DESCRIPTION:
Breast cancer cells are often very dependent on estrogens to continue to grow. Atamestane blocks the formation of estrogens and androgenic precursors in the body. Toremifene blocks circulating and intracellular estrogens from stimulating estrogen receptors in breast cancer cells. The goal of therapy with atamestane, an aromatase inhibitor, in combination with the estrogen receptor antagonist, toremifene, is to achieve maximal suppression of estrogen stimulation of breast cancer cells. This study is designed to determine whether combination therapy will lengthen the time to disease progression and the rate of objective response compared to single agent aromatase inhibitor therapy with letrozole.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 years or older
* Pathological or histological confirmation of breast cancer at initial diagnosis or at the time of metastases
* ECOG performance status of 0, 1 or 2 or Karnofsky performance status of 60 or higher
* Predicted life expectancy of 12 weeks or more
* Postmenopausal endocrine status. LH/FSH levels in the postmenopausal range in women whose menopause occurred less than 5 years ago
* Locally recurrent, locally advanced, locally metastatic disease not amenable to radiation therapy or surgery and/or distant metastatic disease
* At least one tumor localization measurable in 2 dimensions (one diameter at least 2 cm for soft tissue/visceral disease assessed by CT/MRI scan or conventional X-ray technique, one diameter at least 1 cm for bone lesions assessed by conventional X-ray techniques)
* Estrogen receptor and/or progesterone receptor positive (by laboratory/institutional standard) at the time of initial diagnosis or determined during subsequent biopsy/surgery of metastases
* Written informed consent obtained

Exclusion Criteria:

* Prior hormonal therapy to treat locally recurrent, locally advanced or metastatic disease
* Prior adjuvant therapy with aromatase inhibitors or antiestrogens/SERMs within 12 months prior to enrollment
* Progression of disease during therapy with antiestrogens (including SERMs administered for prevention of osteoporosis)
* Life-threatening locally recurrent, locally advanced or metastatic disease or disease requiring chemotherapeutic intervention (such as inflammatory breast cancer)
* History of known CNS metastases, significant neurological dysfunction including active seizures, or clinical signs of other significant neurological diseases
* Other active malignancy (except basal cell carcinoma of the skin or in situ cervical cancer). Patients with previous malignancies must be without evidence of disease for at least five years
* Renal insufficiency (serum creatinine > 2.0 mg/dL)
* Aspartate aminotransferase, alanine aminotransferase or serum bilirubin levels more than 2.5 times upper limit of normal
* Hemoglobin <9 g/dL
* Platelet count of less than 100,000 platelets per mm3
* Total white blood cell count of less than 2,000 cells per mm3
* Premenopausal endocrine status; pregnant or lactating females
* Usage of an investigational drug within the thirty (30) days prior to enrollment; or the planned usage of an investigational drug other than the study medication during the course of the current study
* Contraindication to use of toremifene, atamestane, letrozole or any of the inactive components of their formulations
* Prior enrollment in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 865 (Actual)
Dates: Start 2002-06; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Time to tumor progression | time from randomization to first occurrence of tumor progression, assessed at week 12 and every subsequent 12 weeks for patients continuing in the study for up to approximately 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Goss, M.D., Study Chair — Princess Margaret Hospital, Canada
Locations (63):
- United States (17):
  - Midwest Internal Medicine, PLLC, Lake Havasu City, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - California Cancer Care, Inc., Greenbrae, California
  - Sharp Memorial Hospital, San Diego, California
  - Innovative Medical Research of South Florida Inc., Miami Shores, Florida
  - Georgia Cancer Specialists, Tucker, Georgia
  - Maryland Hematology/Oncology Associates, Baltimore, Maryland
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - Kansas City Oncology and Hematology Group, Kansas City, Missouri
  - Great Falls Clinic-Oncology West, Great Falls, Montana
  - Slocum-Dickson Medical Group, New Hartford, New York
  - Hematology Oncology Consultants, Inc., Columbus, Ohio
  - Oncology Consultants, Houston, Texas
  - First Dynamic Healthcare Services, Inc., Killeen, Texas
  - Cache Valley Cancer Treatment & Research Clinic, Logan, Utah
  - Virginia Oncology Associates, Norfolk, Virginia
  - Western Washington Oncology Inc., P.S., Olympia, Washington
- Canada (4):
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University, Department of Oncology, Montreal, Quebec
- Russia (27):
  - Arkhangelsk Regional Oncology Center, Department of Chemotherapy, Arkhangelsk
  - Tatarstan Republican Clinical Oncology Center, Kazan'
  - Krasnodar Regional Clinical Oncology Center, Chemotherapy Department, Krasnodar
  - Lipetsk Regional Oncology Center, Department of General Oncology, Lipetsk
  - Blokhin Cancer Research Center, Department of Chemotherapy and Combined Treatment of Tumors, Moscow
  - Blokhin Cancer Research Center, Department of Chemotherapy, Moscow
  - Blokhin Cancer Research Center, Department of Clinical Pharmacology and Chemotherapy, Moscow
  - Blokhin Cancer Research Center, Department of New Antitumor Drug Research, Moscow
  - Hertzen Research Institute of Oncology, Department of Chemotherapy, Moscow
  - Central Clinical Hospital of the Ministry of Transport n.a. Semashko, Department of Chemotherapy, Moscow
  - Moscow City Hospital #40, Department of Chemotherapy, Moscow
  - Moscow City Oncology Hospital #62, Moscow
  - Murmansk Regional Oncology Center, Murmansk
  - Municipal Clinical Hospital #1, Department of Breast Tumors, Oncology Department, Novosibirsk
  - Medical Radiological Research Center, Obninsk
  - Ryazan Regional Clinical Oncology Center, Ryazan
  - Leningrad Regional Oncology Center, Saint Petersburg
  - St. Petersburg City Oncology Center, Saint Petersburg
  - Laboratory of Thoracic Oncology, St. Petersburg Pavlov State Medical University, Research Institute of Pulmonology, Saint Petersburg
  - Petrov Research Institute of Oncology, Department of Biotherapy and Bone Marrow Transplantation, Saint Petersburg
  - Petrov Research Institute of Oncology, Department of Breast Cancer, Saint Petersburg
  - Petrov Research Institute of Oncology, Department of Chemotherapy, Saint Petersburg
  - Samara Regional Oncology Center, Department of Chemotherapy, Samara
  - Stavropol Regional Oncology Center, Department of Chemotherapy, Stavropol
  - Research Institute of Oncology, Tomsk Scientific Center, Siberian Department of the Russian Academy of Medical Sciences, Department of Chemotherapy, Tomsk
  - V. Novgorod Regional Oncology Center, Department of Chemotherapy, V. Novgorod
  - Burdenko Voronezh Medical Academy, Oncology Department, Clinical Facility: Regional Clinical Oncology Center, Voronezh
- Ukraine (15):
  - Cherkassy Regional Oncology Center, Chemotherapy Department, Cherkassy
  - Dnepropetrovsk State Medical Academy, Oncology Department. Clinical Facility: Dnepropetrovsk City Clinical Hospital #4, Dnipro
  - Donetsk State Medical University. Clinical Facility: Donetsk Regional Antineoplastic Center, Mammology Department, Donetsk
  - Ivano-Frankovsk State Medical Academy; Oncology Department Clinical Facility: Ivano-Frankovsk Regional Oncology Center, Ivano-Frankivsk
  - Kharkov State Medical University. Clinical Facility: Grigoriev Medical Radiology Institute, Chemotherapy Department, Kharkiv
  - Kharkov Medical Academy of Postgraduate Education, Oncology and Pediatric Oncology Department. Clinical Facility: Kharkov Regional Clinical Oncology Dispensary, Chemotherapy Department, Kharkiv
  - Kiev Central Clinical Hospital, Ukraine Security Services, Surgery Department, Kiev
  - Kiev Oncology Institute, Ukraine Medical Science Academy, Department of Breast Tumors, Kiev
  - Kiev Postgraduate Studies Medical Academy. Clinical Facility: Kiev City Oncology Hospital, Chemotherapy Department, Kiev
  - National Medical University, Oncology Department. Clinical Facility: Kiev City Oncology Hospital, Surgery Department, Kiev
  - Krivoy Rog City Oncology Center, Kryvyi Rih
  - Lviv State Medical University, Oncology and Medical Radiology Department. Clinical Facility: Lviv State Oncology Regional Clinical Diagnostic Center, Chemotherapy Department, Lviv
  - Odessa State Medical University, Oncology Department. Clinical Facility: Odessa Regional Oncology Center, Chemotherapy Department, Odesa
  - Uzhgorod National University Oncology Course of Surgery Department of Postgraduate Education Faculty Clinical Facility: Zakarpatye Regional Oncology Center, Uzhhorod
  - Zaporozhye Statue Institute of Postgraduate Training. Oncology Department; Clinical Facility: Zaporozhye Regional Oncology Center, Zaporizhzhya